CLINICAL TRIAL: NCT04684589
Title: Effect of PDE5 Inhibition on Adipose Metabolism in Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Evan Brittain, Associate Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202420
Record Dates: First submitted 2020-12-16; First posted 2020-12-24 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Tadalafil

STUDY DESIGN:
Intervention Model Description: Half of participants to get tadalafil and half to get placebo.
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tadalafil (Active Comparator): Subjects will be randomized to one of two arms. 50 obese adult subjects will be randomized to the Tadalafil arm following the screening visit. Beginning at their baseline visit, they will receive an oral daily dose of Tadalafil (20mg) that they will take for 12 weeks (through their completion of the study). After randomization has occurred, the active comparator subjects will undergo the following visit protocol: screening visit, baseline visit, an interim visit (10 weeks post-baseline), and a 12-week visit.
  Interventions: Drug: Tadalafil 20 MG
- Placebo (Placebo Comparator): Subjects will be randomized to one of two arms. 50 obese adult subjects will be randomized to the placebo arm following the screening visit. Beginning at their baseline visit, they will receive an oral daily dose of a placebo pill (20mg) that they will take for 12 weeks (through their completion of the study). After randomization has occurred, the placebo comparator subjects will undergo the following visit protocol: screening visit, baseline, an interim visit (10 weeks post-baseline), and a 12-week visit.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil 20 MG — Tadalafil is an FDA approved, clinically-available drug that inhibits the enzyme phosphodiesterase type 5A (PDE5). Subjects who are randomized to this arm will be provided with 20mg of Tadalafil to take every day for 12 weeks, beginning at their baseline visit.
  Other Names: CIALIS
  Arms: Tadalafil
Drug: Placebo — Subjects in this arm will be provided with 20mg Placebo to take every day for 12 weeks, beginning at their baseline visit.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blinded, placebo-controlled study of the effects of PDE5 inhibition with tadalafil on adipose tissue in obese individuals. Adipose metabolism will be measured using magnetic resonance imaging (MRI) scans and by aspirating a small amount of adipose to measure gene expression.

DETAILED DESCRIPTION:
The purpose of this study is to test whether tadalafil causes subcutaneous adipose tissue to have a "beige" phenotype. Participants will be randomized to either placebo or tadalafil for 12 weeks. Investigators will study adipose metabolism using MRI scans and aspiration of subcutaneous adipose from the abdomen. In addition to MRI scans at room temperature, the investigators will use a cooling protocol to test the combined effects of tadalafil and on adipose metabolism. Investigators will also measure the effects of the drug on body composition. In addition to the study visits, participants will wear an activity tracker (Fitbit) and log their dietary intake several times using an online tool. There will be a small amount of radiation exposure. Participants will be compensated for participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Obesity (BMI ≥ 30 kg/m2)

Exclusion Criteria:

* Age <19 or > 50
* BMI < 30 kg/m2
* Systolic blood pressure (SBP) < 100, > 150 mmHg
* Current anti-hypertensive medication use, including diuretics
* Current use of organic nitrates
* Current use of PDE-5 inhibitors (sildenafil, tadalafil, vardenafil)
* History of reaction to PDE-5 inhibitors
* Known HIV infection
* Use of medications that strongly alter CYP3A4 activity
* History of myocardial infarction, angina, uncontrolled cardiac arrhythmia, stroke, transient ischemic attack, or seizure
* Known non-arteritic ischemic optic retinopathy (NAIOR)
* History of hearing loss
* Estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m2 by the modified diet in renal disease (MDRD) equation
* Hepatic transaminase (AST and ALT) levels greater than three times the upper limit of normal
* Known pregnancy or breastfeeding or those unwilling to avoid pregnancy during the course of the study
* History of priapism
* Use in excess of four alcoholic drinks daily
* History of diabetes mellitus or use of anti-diabetic medications
* Known anemia (men, Hct < 38% and women, Hct <36%)
* Menopause
* Weight > 300 pounds
* Individuals with circadian rhythm disorders, shift workers, or those who travel across time zones frequently

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Thermoneutral FSF of WAT at the level of the umbilicus at 12 Weeks. | 12 weeks
  MRI measurement of lipid content
Subcutaneous adipose tissue expression of UCP1 (normalized expression units) | 12 weeks
  Measurement of gene expression in adipose sample

SECONDARY OUTCOMES:
Thermoneutral fat signal fraction of brown adipose tissue | Baseline to 12 weeks
  MRI measurement of lipid content
Cold-exposed fat signal fraction of white adipose tissue and grown adipose tissue | Baseline to 12 weeks
  MRI measurement of lipid content
Subcutaneous adipose tissue gene expression of mitochondrial genes (normalized expression units) | Baseline to 12 weeks
  Measurement of gene expression in adipose sample
Subcutaneous adipose tissue natriuretic peptide receptor expression | Baseline to 12 weeks
  Measurement of gene expression in adipose sample

OTHER OUTCOMES:
BAT perfusion under thermoneutral and cold conditions | Baseline to 12 weeks
  MRI measurement of blood flow
Change in BNP concentration during cold exposure | Baseline to 12 weeks
  Blood measurement of hormone
Change in free fatty acid level during cold exposure | Baseline to 12 weeks
  Blood measurement of fat
Change in whole body subcutaneous and visceral fat mass | Baseline to 12 weeks
  Measurement of fat mass will be examined using dual x-ray absorptiometry to assess for changes in fat mass.
Resting energy expenditure | Baseline to 12 Weeks
  Measurement of energy expended
Homeostatic Index of Insulin Resistance | Baseline to 12 Weeks
  Blood measurement of insulin resistance

CONTACTS AND LOCATIONS:
Overall Officials: Evan Brittain, MD, MSci, Principal Investigator — VUMC
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT04684589/ICF_000.pdf